CLINICAL TRIAL: NCT07123428
Title: A Phase I Clinical Study to Investigate the Safety, Tolerability, and Pharmacokinetics of and Food Effect on TRD205 After Single and Multiple Doses in Healthy Adult Subjects
Brief Title: Single and Multiple Ascending Doses and Food Effect Study of TRD205 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: TRD205-Ⅰ-01
Record Dates: First submitted 2024-01-19; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigator and participant will be masked for the single ascending dose (SAD) study It's open label for multiple ascending dose (MAD) study and group B of food effect study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- TRD205: Single ascending dose (SAD) study (Experimental): TRD205: oral, single ascending doses up to 7 doses levels.
  Interventions: Drug: TRD205
- Placebo: Single ascending dose (SAD) study (Placebo Comparator): Placebo: oral, TRD205 placebo in single ascending doses study.
  Interventions: Drug: Placebo
- TRD205: Food effect study (Experimental): TRD205: oral, just 1 dose under fasted or fed condition for each period.
  Interventions: Drug: TRD205
- Placebo: Food effect study (Placebo Comparator): Placebo: oral, under fasted or fed condition for each period.
  Interventions: Drug: Placebo
- Multiple ascending dose (MAD) study (Experimental): TRD205: oral, multiple ascending doses up to 4 doses levels. Doses and dosing frequency will be decided based on SAD results.
  Interventions: Drug: TRD205

INTERVENTIONS:
Drug: TRD205 — TRD205 tablet
  Arms: Multiple ascending dose (MAD) study; TRD205: Food effect study; TRD205: Single ascending dose (SAD) study
Drug: Placebo — TRD205 placebo tablet
  Arms: Placebo: Food effect study; Placebo: Single ascending dose (SAD) study

SUMMARY:
This is a Phase I clinical study to evaluate the safety, tolerability, and pharmacokinetics of TRD205 after single and multiple doses and to evaluate the effect of food on TRD205 in healthy adult subjects.

DETAILED DESCRIPTION:
This study consists of three parts:

* Single ascending dose study
* Multiple ascending dose study
* Food effect study

ELIGIBILITY:
Inclusion Criteria:

* Subjects who can understand the requirements and potential side effects of the study and voluntarily sign the informed consent form.

  * Able to complete the study per protocol and communicate with the investigators.
  * Subjects (and their sexual partners) should voluntarily practice effective contraception per protocol.
  * Healthy subjects aged 18-55 years.
  * Body weight should be ≥ 50 kg for male subjects and ≥ 45 kg for female subjects with a body mass index of 18-28 kg/m2.
  * Physical examination and vital sign: normal or are considered by the investigator to be of no clinical significance.
  * No vaccination within 30 days prior to screening.

Exclusion Criteria:

* Smoking 5 or more cigarettes per day within 3 months before screening.
* Subjects with an allergic constitution, such as a history of allergy to two or more drugs or food.
* Subjects who have a history of drug abuse and or alcoholism.
* Subjects who have had blood donation and/or blood loss ≥ 450 mL wihin 3 months before screening.
* Subjects who have consumed medications known to alter hepatic drug metabolism enzyme activity within 28 days before screening.
* Subjects who have taken any other prescription medication, OTC products, vitamins or herbal products within 14 days before screening, except for those exempted by the investigator on a case-by-case basis.
* Subjects who have eaten special food, such as dragon fruit, mango, pomelo, grapefruit, cranberry and their juice, or had vigorous exercise, or had other factors that may influence the ADME process of drug.
* Subjects who have concomitant drugs that induce or inhibit CYP3A4, P-gp, Bcrp.
* Subjects who have consumed investigational products or participated in drug clinical trials within 3 months before taking IP.
* Subjects who have dysphagia or other gastrointestinal diseases that can influence drug adsorption.
* Subjects who can not tolerate the standard meal (just for those who participate the food effect study).
* 12-lead ECG: abnormal results and considered by the investigator to be of clinical significance.
* Pregnant or lactating women.
* Laboratory tests: abnormal results and considered by the investigator to be of clinical significance. Or subjects with the diseases of gastrointestinal tract, kidney, liver, nervous system, blood system, endocrinal system, tumor, lung, immunity, mental system, cardiovascular system, cerebral vascular system within 12 months before screening.
* Positive serological tests for hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), and treponema pallidum (TP) at screening.
* Subjects who have had acute disease or concomitant drugs from screening to taking IP.
* Subjects who have consumed chocolate, Caffeine-containing products or xanthine containing food (such as tea, coffee, colar) within 48 hours beforing taking IP.
* Subjects who have consumed alcohol-containing products within 48 hours beforing taking IP.
* Subjects who have a positive urine drug screening test result.
* Subject who have received surgery within 4 weeks before taking IP.
* Subject who are not ready to abstain from participation in any other clinical study for the duration of this study and for 30 days or more (as required by the investigator) after completion of the study.
* Mental or physical disability.
* Subject cannot tolerate venipuncture blood collection or has a history of sickness at the sight of blood and/or needle.
* Any reason that, in the opinion of the Investigator, may prevent the subject from participating in the study.
* Subjects who have the risk factors of torsade de pointes, or a family history of a first-degree relative with short QT syndrome, long QT syndrome, unexplained sudden death in youth, drowning, or sudden infant death syndrome.
* Subjects with abnormal and clinically significant hyperkalemia, hypokalemia, hypermagnesemia, hypomagnesemia, hypercalcemia or hypocalcemia as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 151 (Actual)
Dates: Start 2024-01-26 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Treatment-Related Adverse Events | After a single dose and/or once daily for 10 consecutive doses
  The safety and tolerability of TRD205 orally administered once and/or multiple times on an empty stomach in healthy subjects

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve （AUC） | After a single dose and/or once daily for 10 consecutive doses
  To evaluate the pharmacokinetic characteristics of a single oral administration of TRD205 in healthy subjects on an empty stomach; To evaluate the pharmacokinetic characteristics of TRD205 orally administered multiple times in healthy subjects; Explore the impact of food on in vivo exposure to TRD205.
Peak Plasma Concentration（Cmax） | After a single dose and/or once daily for 10 consecutive doses
  To evaluate the pharmacokinetic characteristics of a single oral administration of TRD205 in healthy subjects on an empty stomach; To evaluate the pharmacokinetic characteristics of TRD205 orally administered multiple times in healthy subjects; Explore the impact of food on in vivo exposure to TRD205.
time to peak（Tmax） | After a single dose and/or once daily for 10 consecutive doses
  To evaluate the pharmacokinetic characteristics of a single oral administration of TRD205 in healthy subjects on an empty stomach; To evaluate the pharmacokinetic characteristics of TRD205 orally administered multiple times in healthy subjects; Explore the impact of food on in vivo exposure to TRD205.
Elimination rate constant（Kel） | After a single dose and/or once daily for 10 consecutive doses
  To evaluate the pharmacokinetic characteristics of a single oral administration of TRD205 in healthy subjects on an empty stomach; To evaluate the pharmacokinetic characteristics of TRD205 orally administered multiple times in healthy subjects; Explore the impact of food on in vivo exposure to TRD205.
apparent volume of distribution（Vd） | After a single dose and/or once daily for 10 consecutive doses
  To evaluate the pharmacokinetic characteristics of a single oral administration of TRD205 in healthy subjects on an empty stomach; To evaluate the pharmacokinetic characteristics of TRD205 orally administered multiple times in healthy subjects; Explore the impact of food on in vivo exposure to TRD205.
elimination half life（T1/2） | After a single dose and/or once daily for 10 consecutive doses
  To evaluate the pharmacokinetic characteristics of a single oral administration of TRD205 in healthy subjects on an empty stomach; To evaluate the pharmacokinetic characteristics of TRD205 orally administered multiple times in healthy subjects; Explore the impact of food on in vivo exposure to TRD205.
Mean retention time（MRT） | After a single dose and/or once daily for 10 consecutive doses
  To evaluate the pharmacokinetic characteristics of a single oral administration of TRD205 in healthy subjects on an empty stomach; To evaluate the pharmacokinetic characteristics of TRD205 orally administered multiple times in healthy subjects; Explore the impact of food on in vivo exposure to TRD205.

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No